CLINICAL TRIAL: NCT03980730
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Studies to Evaluate the Safety and Efficacy of Azeliragon as a Treatment for Subjects With Mild Alzheimer's Disease and Impaired Glucose Tolerance
Brief Title: Study of Azeliragon in Patients With Mild Alzheimer's Disease and Impaired Glucose Tolerance
Acronym: Elevage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: for business reasons
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTP488-305
Record Dates: First submitted 2019-05-31; First posted 2019-06-10 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer Disease
Keywords: Receptor for Advanced Glycation Endproducts (RAGE); ADAS-cog; CDR-sb
MeSH Terms: conditions — Alzheimer Disease | interventions — azeliragon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azeliragon (Experimental): Azeliragon 5mg capsule administered orally, once daily for 6 months (Part 1) or 18 months (Part 2)
  Interventions: Drug: Azeliragon
- Placebo (Placebo Comparator): Matching placebo capsule administered orally, once daily for 6 months (Part 1) or 18 months (Part 2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azeliragon — Azeliragon 5 mg capsule administered orally, once daily
  Other Names: TTP488
  Arms: Azeliragon
Drug: Placebo — Matching placebo capsule administered orally, once daily
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of azeliragon in patients with mild Alzheimer's disease and impaired glucose tolerance. Patients will receive either azeliragon or placebo with a patient's participation lasting approximately 9 months (in Part 1) or 21 months (in Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer Disease (AD) with documented evidence of progression of disease
* Mini Mental State Examination (MMSE) score of 21-26, inclusive
* Clinical Dementia Rating global score of 0.5 or 1
* Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog14) of 10 or more
* Brain magnetic resonance imaging (MRI) consistent with the diagnosis of probable AD
* Concurrent use of cholinesterase inhibitor or memantine with stable dose for at least 2 months prior to screening
* Hemoglobin A1c (HbA1c) 6.5% - 9.5%, inclusive
* Caregiver willing to participate and be able to attend clinic visits with patient
* Ability to ingest oral medications

Exclusion Criteria:

* Significant neurological or psychiatric disease other than Alzheimer's disease
* Previous clinical trial participation within 90 days of screening
* Previous exposure to putative disease modifying therapy for Alzheimer's disease within 1 year of screening
* History of cancer within the last 5 years except adequately treated cervical carcinoma in-situ, cutaneous basal cell or squamous cell cancer, or non-progressive prostate cancer not requiring current treatment
* Women of childbearing potential
* Uncontrolled blood pressure and/or blood pressure above 140/90
* Participants receiving medications that may negatively impact cognitive function
* History of diabetic ketoacidosis within the past year
* History of chronic pancreatitis
* Stage 4 kidney disease
* Use of insulin therapy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (27):
  - Tucson Neuroscience Research, Tucson, Arizona
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Charter Research, Lady Lake, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - ClinCloud, Maitland, Florida
  - Synexus Clinical Research US, Orlando, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - The Roskamp Institute, Sarasota, Florida
  - Brain Matters Research, Stuart, Florida
  - Emory Alzheimer's Clinical Research Unit, Atlanta, Georgia
  - NeuroStudies.net LLC, Decatur, Georgia
  - IU Health Partners, Adult Neurology Clinic, Indianapolis, Indiana
  - Memory Center / Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millennium Psychiatric Associates, St Louis, Missouri
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Clarity Clinical Research, East Syracuse, New York
  - Neurological Associates of Long Island, Lake Success, New York
  - ANI Neurology dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Summit Research Network, Portland, Oregon
  - Center for Cognitive Health, Portland, Oregon
- Canada (6):
  - Okanagan Clinical Trials Ltd., Kelowna, British Columbia
  - True North Clinical Research Inc., Halifax, Nova Scotia
  - True North Clinical Research Inc., Kentville, Nova Scotia
  - Recherches Neuro-Hippocampe, Ottawa, Ontario
  - Recherches Neuro-Hippocampe Inc., Gatineau, Quebec
  - Q&T Research Sherbrooke Inc, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azeliragon: Azeliragon 5mg capsule administered orally, once daily for 6 months (Part 1)
  Azeliragon: Azeliragon 5 mg capsule administered orally, once daily
- Placebo: Matching placebo capsule administered orally, once daily for 6 months (Part 1)
  Placebo: Matching placebo capsule administered orally, once daily
Period: Overall Study
Arm/Group | Azeliragon | Placebo
Started | 21 | 22
Completed | 19 | 18
Not Completed | 2 | 4
Not completed — Study Terminated by Sponsor | 0 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Sponsor Request | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azeliragon | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (5.82) | 77.0 (6.56) | 76.7 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years Since Diagnosis of AD [Mean (Standard Deviation); unit: years] | 1.9 (1.16) | 1.8 (1.24) | 1.9 (1.19)
Education Level [Count of Participants; unit: Participants]
  Some College | 5 | 2 | 7
  Other (Training, Certifications, etc.) | 1 | 2 | 3
  Master's Degree | 1 | 4 | 5
  High School | 6 | 8 | 14
  Associate's Degree | 1 | 2 | 3
  Bachelor's Degree | 7 | 4 | 11
ApoE4 Carrier Status [Count of Participants; unit: Participants]
  Non-Carrier | 9 | 12 | 21
  Carrier | 12 | 10 | 22
ADAS-Cog 14 Total Score [Mean (Standard Deviation); unit: units on a scale] — The Alzheimer's Disease Assessment Scale - Cognitive Subscale 14 Item (ADAS-cog14) scoring range is from 0 to 90, with higher scores indicating greater cognitive impairment
  units on a scale | 30.8 (7.53) | 29.4 (8.87) | 30.1 (8.17)
CDR Global Score [Count of Participants; unit: Participants] — Clinical Dementia Rating global scores are 0 for cognitively unimpaired individuals, 0.5 for questionable dementia, 1 for mild dementia, 2 for moderate dementia and 3 for severe dementia.
  Participants
    CDR Global = 1 | 11 | 9 | 20
    CDR Global = 0.5 | 10 | 13 | 23
CDR Sum of Boxes [Mean (Standard Deviation); unit: units on a scale] — Clinical Dementia Rating - Sum of box (CDR-sb) scores range from 0 to 18 with higher scores indicating greater cognitive impairment
  units on a scale | 4.7 (1.37) | 4.2 (2.22) | 4.5 (1.85)
MMSE Total Score [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Exam scale range is 0 to 30 with lower scores indicating greater cognitive impairment.
  units on a scale | 23.7 (1.48) | 23.5 (2.24) | 23.6 (1.89)

OUTCOME MEASURES:

1. Primary Outcome: Part 1 : Change From Baseline in the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog14) at Month 6
Description: The Alzheimer's Disease Assessment Scale - Cognitive Subscale 14 Item (ADAS-cog14) scoring range is from 0 to 90, with higher scores indicating greater cognitive impairment
Time Frame: Baseline to Month 6
Population: The full analysis set (FAS) includes all randomized subjects, whether or not they receive any study medication, and who have at least one post-Baseline assessment. The FAS was used for all hypothesis tests of efficacy.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Azeliragon | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale | 1.8 (0.82) | 0.4 (0.69)
Statistical Analysis 1: Comparison: Azeliragon vs Placebo; Test type: Superiority; p = 0.2057, Mixed Models Analysis

2. Secondary Outcome: Part 1: Change From Baseline in the Amsterdam-Instrumental Activities of Daily Living (Amsterdam-IADL) at Month 6
Description: The Amsterdam-Instrumental Activities of Daily Living score is calculated from a questionnaire consisting of 70 items in seven categories using an item response theory method of scoring. Scores range from 20 to 80 where lower scores indicate greater functional impairment.
Time Frame: Baseline to Month 6
Population: The full analysis set (FAS) includes all randomized subjects, whether or not they receive any study medication, and who have at least one post-Baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Azeliragon | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale | 6.2 (1.99) | 9.3 (2.37)

3. Secondary Outcome: Part 1: Change From Baseline in the Clinical Dementia Rating Scale-Sum of Boxes (CDR-sb) at Month 6
Description: Clinical Dementia Rating - Sum of box (CDR-sb) scores range from 0 to 18 with higher scores indicating greater cognitive impairment.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Azeliragon | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale | 0.6 (0.29) | 1.3 (0.36)

4. Secondary Outcome: Part 1: Change From Baseline in the Functional Activities Questionnaire (FAQ) at Month 6
Description: The total FAQ score ranges from 0 to 30, with higher scores indicating greater functional loss.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Azeliragon | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale | -0.5 (0.84) | 2.8 (0.84)

5. Secondary Outcome: Mean Change From Baseline in the Mini Mental State Exam (MMSE) at Month 6.
Description: The MMSE scale range is 0 to 30 with lower scores indicating greater cognitive impairment.
Time Frame: Baseline to Month 6
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Azeliragon | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale | -1.8 (0.41) | -1.7 (0.43)

6. Other Pre Specified Outcome: Count and Percentage of Subjects With Treatment-emergent Adverse Events
Time Frame: Baseline to Month 6
Population: The safety set (SAF) includes all subjects who receive any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Azeliragon | Placebo
Number analyzed (Participants) | 21 | 22
Participants
  Subjects with at least 1 adverse event | 16 | 16
  Subjects with at least 1 serious adverse event | 1 | 0
  Subjects who had drug withdrawn due to AE | 2 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Azeliragon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22
Other Adverse Events (participants affected / at risk) | 9/21 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azeliragon (N=21) | Placebo (N=22)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azeliragon (N=21) | Placebo (N=22)
Urinary tract infection (Infections and infestations) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Where PI requires the use of the Study Results for publication, the PI shall seek the Sponsor's written approval which shall not be unreasonably withheld; provided, however, that (i) Sponsor may require removal of any Confidential Information of Sponsor or may delay publication for a reasonable period of time in order to secure protection any IP Rights; and, (ii) as the Study is designed as a multi-center Study, no publication shall be made until after the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03980730/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT03980730/SAP_001.pdf